CLINICAL TRIAL: NCT06006208
Title: Ventilation During Intensive Care Unit Transport After Cardiac Surgeries; When Should we Use a Ventilator?
Brief Title: AMBU Bag Manual Ventilation vs. Transport Ventilator Mechanical Ventilation for Transport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Yoshihisa Morita, MD, Associate professor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: iRISID-2022-1315
Record Dates: First submitted 2023-08-06; First posted 2023-08-23 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Oxygenation; Manual Ventilation; Mechanical Ventilation; Point of Care Ultrasound; Cardiac Function Disturbance Postoperative
Keywords: ventilator; point of care ultrasound; transport

STUDY DESIGN:
Intervention Model Description: After IRB approval and obtaining a written informed consent, patients will be randomly assigned to the one of the following 2 arms. However, AMBU bag arm patients may be switched to Hamilton C1 at an anesthesia provider's discretion based on post cardiopulmonary bypass right ventricular function, PaO2/FiO2, and PaCO2. These patients will be excluded from the AMBU bag arm.
  Arm 1: AMBU bag manual ventilation during transport to the ICU Arm 2: Hamilton C1 ventilator during transport to the ICU
Who Masked: Participant
Masking Description: The patients will be randomly assigned to 2 arms above and the patients are not informed about which arm they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1: AMBU bag manual ventilation during transport to the ICU (No Intervention)
- Arm 2: Hamilton C1 ventilator during transport to the ICU (Experimental)
  Interventions: Device: Hamilton C1 ventilator during transport to the ICU

INTERVENTIONS:
Device: Hamilton C1 ventilator during transport to the ICU — Instead of AMBU bag manual ventilation during transport to the ICU, intervention is using Hamilton C1 ventilator during transport to the ICU
  Arms: Arm 2: Hamilton C1 ventilator during transport to the ICU

SUMMARY:
This is a clinical trial to compare the oxygenation and ventilation performance between manual ventilation and mechanical ventilation when transporting cardiac patients to the ICU.

DETAILED DESCRIPTION:
Following cardiac surgery, patients often require ventilation during transport to the intensive care unit (ICU). Most of the time, manual ventilation using an AMBU bag (AMBU INC. MD, USA) is utilized, but some patients need mechanical ventilation due to concern for oxygenation, ventilation, and hemodynamics. The indication to choose mechanical ventilation over manual ventilation is determined on a case-by-case basis, mostly based on providers' experiences or surgical request, because currently there is no clear clinical evidence behind that. With this clinical study, the investigators intend to build up clinical evidence by comparing oxygenation, ventilation, hemodynamics, and cardiac functions between two arms: manual ventilation using AMBU bag arm and mechanical ventilation using a transport ventilator.

Objective: In this study, the investigators plan to compare the effects of transport ventilators (Hamilton C1: Bodaduz, Schweiz) and AMBU bag manual ventilation on oxygenation, ventilation, biventricular function, and hemodynamics. This is a two-arm study.

1. To assess pre and post transport PaO2/FiO2 (P/F ratio), PaCO2, biventricular function, and mean artery pressure in the AMBU bag and Hamilton transport ventilator groups. The investigators hypothesize that using the Hamilton transport ventilator will show a smaller change in P/F ratio, mean artery blood pressures and biventricular function compared to the AMBU bag group. If true, these findings would support using the Hamilton ventilator for transport in appropriate surgical patients.
2. To perform "in-vitro" flow analysis using a flow analyzer analyzer (CITREX H5:

Buchs, Schweiz) and lung simulator (SmartLung 2000: Buchs, Schweiz) to measure the accuracy of the ventilations of Hamilton C1 ventilator and AMBU bag manual ventilation on different resistance and compliance settings of the lung simulator

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old (any gender or race)
* Cardiac surgery
* Require postoperative mechanical ventilation and care in the ICU.

Exclusion Criteria:

* Patients' refusal
* Extubation in OR
* On mechanical circulatory support
* Requirement for postoperative therapy with inhaled pulmonary vasodilators (epoprostenol (FLOLAN), inhaled nitric oxide, etc.)
* Severe RV dysfunction with preoperative echocardiography
* Contraindication to TEE and pulmonary artery catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment was done from November 1, 2023, to October 9, 2024. Location was a university medical center. Patients aged > 18 years who underwent full sternotomy cardiac surgery and required postoperative ICU care were included in the study. The exclusion criteria included extubation in the operating room, postoperative need for mechanical circulatory support, postoperative open chest, and continuous inhalation of epoprostenol or nitric oxide.
Pre-assignment Details: Patients who needed to be switched the ventilation method from the originally designated method were excluded from the study before assignment to the arms.
Groups:
- Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU: patients who were transported to the ICU with manual (AMBU bag) ventilation
- Arm 2: Hamilton C1 Ventilator During Transport to the ICU: patients who were transported to the ICU with mechanical (Hamilton C1) ventilation
Period: Overall Study
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
Started | 39 | 39
Completed | 38 | 39
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years old] | 61.42 (130.8) | 66.92 (8.83) | 64.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 25 | 29 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 29 | 38 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: The % Changes in PaO2/FiO2 (P/F Ratio)
Description: The % changes in PaO2/FiO2 (P/F ratio) pre and post transport to ICU. P/F ratio will be assessed on arterial blood gas immediately before and after the transport to ICU, at the same time as the investigators do echocardiographic assessment as described above.
  i.e. (post-transport measurement - pre-transport measurement)/pre-transport measurement x100 (%)
Time Frame: First aortic blood gas analysis Immediately before transport to ICU till the second arterial blood gas analysis after dropping off the patient at ICU; approximately 30 minutes after the first visual assessment.
Measure: Median (Inter-Quartile Range); unit: The percent change in PF ratio
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
Number analyzed (Participants) | 38 | 39
The percent change in PF ratio | 6.76 [-18.61 to 36.26] | -12.2 [-38.56 to 17.94]
Statistical Analysis 1: Comparison: Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU vs Arm 2: Hamilton C1 Ventilator During Transport to the ICU; Test type: Superiority; p = 0.275, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The % Change in PaCO2
Description: The % changes in PaCO2 pre and post transport to ICU. PaCO2 will be assessed on arterial blood gas immediately before and after the transport to ICU, at the same time as the investigators do echocardiographic assessment as described above.
  i.e. (post-transport measurement - pre-transport measurement)/pre-transport measurement x100 (%)
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: The percent change in PaCO2
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
Number analyzed (Participants) | 38 | 39
The percent change in PaCO2 | 3.42 [-10.0 to 9.08] | 3.06 [-8.46 to 11.31]
Statistical Analysis 1: Comparison: Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU vs Arm 2: Hamilton C1 Ventilator During Transport to the ICU; Test type: Superiority; p = 0.891, Wilcoxon (Mann-Whitney)

3. Primary Outcome: The % Change in Mean Artery Blood Pressure
Description: The % change in mean artery blood pressure before and after the transport to the ICU.
  i.e. (post-transport measurement - pre-transport measurement)/pre-transport measurement x100 (%)
Time Frame: Pre-transport hemodynamic values were averaged from the final three readings (taken at 1-min intervals) before switching to the transport monitor, and post-transport readings were recorded immediately after transfer to the ICU monitor.
Measure: Mean (Standard Deviation); unit: % change in mean artery pressure
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
Number analyzed (Participants) | 38 | 39
% change in mean artery pressure | -3.73 (18.04) | 13 (15.61)

4. Secondary Outcome: The Visual Scale in Changes in Left Ventricular Function
Description: Within-group and between-group changes in visual assessment of left ventricular function parameters before and after transport (1: severe hypokinetic, 2: moderate hypokinetic, 3: mild hypokinetic, 4: normal, 5: hyperdynamic)
Time Frame: First visual assessment of left ventricular function Immediately before transport to ICU till the second visual assessment after dropping off the patient at ICU; approximately 30 minutes after the first visual assessment.
Population: The number of participants who had a change in visual assessment of left ventricular function pre and post-transport
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
Number analyzed (Participants) | 38 | 39
Participants | 0 | 0

5. Secondary Outcome: The Visual Scale in Changes in Right Ventricular Function
Description: Within-group and between-group changes in visual assessment of right ventricular cardiac function parameters before and after transport (1: severe hypokinetic, 2: moderate hypokinetic, 3: mild hypokinetic, 4: normal, 5: hyperdynamic)
Time Frame: First visual assessment of right ventricular function Immediately before transport to ICU till the second visual assessment after dropping off the patient at ICU; approximately 30 minutes after the first visual assessment.
Population: The number of participants who had a change in visual assessment of right ventricular function pre and post-transport
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
Number analyzed (Participants) | 38 | 39
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 12 weeks
Arm/Group | Arm 1: AMBU Bag Manual Ventilation During Transport to the ICU | Arm 2: Hamilton C1 Ventilator During Transport to the ICU
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT06006208/Prot_SAP_ICF_002.pdf